CLINICAL TRIAL: NCT01363505
Title: Is Intravesicular Pressure a Better Tool to Predict Renal Failure in Critically Ill Patients Compared With Routine Hemodynamic Parameters?
Brief Title: Bladder Pressure Predicting Renal Failure in Critically Ill Patients as Compared to Hemodynamic Parameters
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Nephrology Attending, Assoc. Chair of Medicine, Northwell Health
Other Study IDs: 11-021
Record Dates: First submitted 2011-05-24; First posted 2011-06-01 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Acute Heart Failure; Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute CHF patients: Acute CHF patients with BARD Intra-abdominal pressure monitors in ICU
  Interventions: Device: BARD® Intra-abdominal Pressure monitor

INTERVENTIONS:
Device: BARD® Intra-abdominal Pressure monitor — monitor linked to foley catheter that is able to measure pressure inside bladder

SUMMARY:
Studies have shown that more than 30% of the overall acute decompensated heart failure (ADHF) patients develop renal dysfunction.

Several studies have tried to find a correlation between hemodynamic Parameters (blood pressure , heart rate, central venous pressure CVP) and worsening of renal function in acute decompensated heart failure patients.

Results showed that there were no correlation between baseline hemodynamics or change in hemodynamics and worsening of renal function.

Another study showed that intra-abdominal pressure (IAP) measuring was a better corollary to renal failure status then measuring cardiovascular hemodynamics using pulmonary artery catheterization in ADHF patients.. An increased IAP was associated with worse renal function and that level of IAP far below abdominal compartment syndrome may adversely affect renal function in patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Any ICU(intensive care unit) or CCU(critical care unit) patient older than 18 y.
* Patient diagnosed on admission with pulmonary edema/CHF (fluid in the lungs) - independently from the baseline renal function.
* No subject will be accepted to take part in the study unless they are able to sign or if Health care proxy signs a consent

Exclusion Criteria:

* Pregnant women
* Cognitively impaired patients
* Age<18 yrs old
* Patients diagnosed on admission with ARDS.
* Patients admitted with a diagnosis of sepsis ( WBC> 12000, CXR findings consistent with pneumonia, positive blood cultures on admission, UTI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied group will consist of patients admitted to the ICU (intensive care unit) or CCU(coronary care ubnit) with evidence of ADHF. We aim in our study to find out if there is a linear relationship between worsening of renal function , IAP ,hemodynamic (CVP) and blood chemical measurements
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
High intraabdominal pressure and effect on renal function | from admission (baseline) until 72 hours later
  IAP measurements will be recorded concomitantly with renal indices. Correlations will be made in regard to pressure measurements and worsening renal function.

SECONDARY OUTCOMES:
Effect of diuretics use on intrabdominal pressure | 3 days from admission
  Early initiation of diuretics in acute heart failure improvement correlating with decreasing IAP measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Study Director — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Background] Cheatham ML, Malbrain ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. II. Recommendations. Intensive Care Med. 2007 Jun;33(6):951-62. doi: 10.1007/s00134-007-0592-4. Epub 2007 Mar 22. PMID 17377769
- [Background] Cheatham ML, Safcsak K. Intraabdominal pressure: a revised method for measurement. J Am Coll Surg. 1998 May;186(5):594-5. doi: 10.1016/s1072-7515(98)00122-7. No abstract available. PMID 9583702
- [Background] Geisberg C, Butler J. Addressing the challenges of cardiorenal syndrome. Cleve Clin J Med. 2006 May;73(5):485-91. doi: 10.3949/ccjm.73.5.485. PMID 16708717